CLINICAL TRIAL: NCT02155309
Title: Pharmacokinetic and Efficacy Profile of Low-Dose Intranasal Scopolamine Spray for Motion Sickness
Brief Title: Pharmacokinetic and Efficacy Profile Intranasal Scopolamine Spray
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Business reason
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAMRUD.2013.0004
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Motion Sickness
Keywords: scopolamine; motion; sickness
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scopolamine (Experimental): 0.2 mg intranasal scopolamine, single dose
  Interventions: Drug: Scopolamine
- Placebo (Placebo Comparator): placebo intranasal (0.1 mg per nostril), single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Scopolamine
  Arms: Scopolamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Part 1, the pharmacokinetic (PK) phase, will expand upon the pilot study conducted at Naval Medical Research Laboratory (NAMRL) and has the goal of determining bioavailability and time to Cmax in a larger representative sample. Part 2, the efficacy phase, is to determine the efficacy of the aqueous spray solution via exposure to a nausea-inducing stimulus.

DETAILED DESCRIPTION:
Part 1: The pharmacokinetic (PK) phase Objective: To determine the bioavailability and amount of scopolamine absorbed after administration of 0.2 mg intranasal scopolamine at regular intervals across 8 hours post- dose.

Hypothesis: Detectable levels of Intranasal scopolamine (INSCOP) will be present in subject plasma within 15 minutes post-dose; mean time to Cmax (maximum plasma concentration) will be less than 1.5 hr.

Part 2: The Efficacy phase Objective: To determine the effectiveness, cognitive performance effects, and medication side-effect profile of 0.2 mg intranasal scopolamine spray as a motion sickness (MS) countermeasure.

Hypothesis: The primary hypothesis is that the INSCOP spray will be more efficacious against MS than placebo, without statistically significant cognitive performance side-effects. Specifically, participants will tolerate significantly more provocative head tilts in the INSCOP condition than in the placebo condition.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 to 59 years old, inclusive, in good general health as determined by physical examination and without clinically significant laboratory profiles
* Normal weight for body size, based on Physical Readiness Test Body Composition Assessment (PPRTBCA) table
* Willing and able to comply with study requirements and restrictions; and read and sign the informed consent.

Exclusion Criteria:

* Known and/or documented drug allergies, especially to scopolamine
* Use of an investigational drug within 30 days of starting the study
* Smoking or use of tobacco products, including "chew" or "snuff", within six months
* Blood donation or significant blood loss within 30 days of starting the study
* Significant gastrointestinal disorder, asthma, or seizure disorders
* History of narrow-angle glaucoma
* History of urinary retention problems
* History of alcohol or other drug abuse
* Pregnancy or suspected pregnancy, or lactation
* Hematocrit values less than 41% for males and 37% for females
* Recent nasal, nasal sinus or nasal mucosa surgery
* Use of prescription, over-the-counter, or herbal medication in past 7 days

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willliam J Becker, Phd, Principal Investigator — Naval Medical Research Unit - Dayton
Locations (1):
- Naval Medical Research Unit, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klocker N, Hanschke W, Toussaint S, Verse T. Scopolamine nasal spray in motion sickness: a randomised, controlled, and crossover study for the comparison of two scopolamine nasal sprays with oral dimenhydrinate and placebo. Eur J Pharm Sci. 2001 May;13(2):227-32. doi: 10.1016/s0928-0987(01)00107-5. PMID 11297908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled subjects who were active-duty military or reserves on active duty status between the ages of 18 and 59 from the Wright-Patterson Air Force Base located in Dayton, Ohio. The last subjects completed in August 2015.
Pre-assignment Details: For the Pharmacokinetics part, 21 subjects were screened, and 13 completed the pharmacokinetics portion. For Efficacy, 42 subjects were screened, and 23 completed, with one removed from efficacy tabulated results due to noncompliance with study protocol. All subjects randomized into treatment order with cross-over design.
Groups:
- PK: Scopolamine Only, Open-label: Baseline vitals, blood draw, and cognitive testing applied. Subjects then received one dose of 0.2 mg intranasal scopolamine (0.1 mg per nostril). No placebo or efficacy. Blood draws, vitals collection, cognitive testing, and subjective fatigue collected for approximately eight hours post-dose.
- Efficacy: Scopolamine, Then Placebo: Subjects received one dose of 0.2 mg intranasal scopolamine (0.1 mg per nostril) for the first of two Efficacy sessions, and then one dose of 0.2 mg placebo intranasal (0.1 mg per nostril) for the second Efficacy session. A minimum of one week separated the two sessions. Each session was identical except for contents of intranasal spray. Baseline vitals, blood draw, and cognitive testing applied prior to dosage. Approximately 40 minutes post-dose, subjects experience mechanical rotation via Coriolis cross-coupling in a stairwise progression until subject reported either full minute of unabated stomach awareness, or the maximum rotation of 40 rpm obtained. Blood draws, vitals collection, cognitive testing and subjective fatigue collected for approximately three hours post-rotation.
- Efficacy: Placebo, Then Scopolamine: Subjects received one dose of 0.2 mg intranasal placebo (0.1 mg per nostril) for the first of two Efficacy sessions, and then one dose of 0.2 mg intranasal scopolamine (0.1 mg per nostril) for the second Efficacy session. A minimum of one week separated the two sessions. Each session was identical except for contents of intranasal spray. Baseline vitals, blood draw, and cognitive testing applied prior to dosage. Approximately 40 minutes post-dose, subjects experience mechanical rotation via Coriolis cross-coupling in a stairwise progression until subject reported either full minute of unabated stomach awareness, or the maximum rotation of 40 rpm obtained. Blood draws, vitals collection, cognitive testing and subjective fatigue collected for approximately three hours post-rotation.
Period: Overall Study
Arm/Group | PK: Scopolamine Only, Open-label | Efficacy: Scopolamine, Then Placebo | Efficacy: Placebo, Then Scopolamine
Started | 13 | 10 | 13
Completed | 13 | 10 | 12
Not Completed | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Efficacy: All Study Participants (Crossover, Double-Blind): Double-blind, placebo-controlled, cross-over design. Study medications (0.2 mg of intranasal scopolamine and 0.2 mg of intranasal placebo) were randomized, blinded, and delivered in identical containers. Each subject participated in two sessions separated by minimum of one week, each session identical except for contents of intranasal spray. Order of treatment and placebo administration randomized. Baseline vitals, blood draw, and cognitive testing applied prior to dosage. Approximately 40 minutes post-dose, subjects experience mechanical rotation via Coriolis cross-coupling in a stairwise progression until subject reported either full minute of unabated stomach awareness, or the maximum rotation of 40 rpm obtained. Blood draws, vitals collection, cognitive testing and subjective fatigue collected for approximately three hours post-rotation.
- Total: Total of all reporting groups
Arm/Group | PK: Scopolamine Only, Open-label | Efficacy: All Study Participants (Crossover, Double-Blind) | Total
Number analyzed (Participants) | 13 | 23 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 23 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.31 (12.59) | 30.96 (10.86) | 30.72 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject was not analyzed due to protocol noncompliance.
  Participants
    number analyzed (Participants) | 13 | 22 | 35
    Female | 3 | 5 | 8
    Male | 10 | 17 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 23 | 36

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Number of Head Movements During Rotation
Description: During rotation, efficacy is measured by the number of head movements subjects are able to make (12 per minute). While seated yaw-axis rotating, a pre-recorded computerized voice informed subjects to make paced head tilts of 30 ̊ to the right and left at a rate of 0.125 Hz (right, center, left, and back to center over 16 seconds).
Time Frame: 40 min
Measure: Mean (Standard Deviation); unit: Number of head tilts
Groups:
- Efficacy: Scopolamine and Placebo (Crossover, Double-blind): Subjects received either one dose of 0.2 mg intranasal scopolamine (0.1 mg per nostril) or one dose of 0.2 mg placebo intranasal (0.1 mg per nostril) for two Efficacy sessions. Each session identical except for contents of intranasal spray. Baseline vitals, blood draw, and cognitive testing applied prior to dosage. Approximately 40 minutes post-dose, subjects experience mechanical rotation via Coriolis cross-coupling in a stairwise progression until subject reported either full minute of unabated stomach awareness, or the maximum rotation of 40 rpm obtained. Blood draws, vitals collection, cognitive testing and subjective fatigue collected for approximately three hours post-rotation. One week minimum separated the two Efficacy sessions.
Arm/Group | PK: Scopolamine Only, Open-label | Efficacy: Scopolamine and Placebo (Crossover, Double-blind)
Number analyzed (Participants) | 0 | 22
Number of head tilts
  Head Tilts: Scopolamine Condition |  | 222.5 (105)
  Head Tilts: Placebo Condition |  | 191.7 (95.1)

ADVERSE EVENTS:
Groups:
- Efficacy: Scopolamine (Crossover, Double-blind); Efficacy: Placebo (Crossover, Double-blind): Subjects received either one dose of 0.2 mg intranasal scopolamine (0.1 mg per nostril) or one dose of 0.2 mg placebo intranasal (0.1 mg per nostril) for two Efficacy sessions. Each session identical except for contents of intranasal spray. Baseline vitals, blood draw, and cognitive testing applied prior to dosage. Approximately 40 minutes post-dose, subjects experience mechanical rotation via Coriolis cross-coupling in a stairwise progression until subject reported either full minute of unabated stomach awareness, or the maximum rotation of 40 rpm obtained. Blood draws, vitals collection, cognitive testing and subjective fatigue collected for approximately three hours post-rotation. One week minimum separated the two Efficacy sessions.
Arm/Group | PK: Scopolamine Only, Open-label | Efficacy: Scopolamine (Crossover, Double-blind) | Efficacy: Placebo (Crossover, Double-blind)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 11/13 | 18/23 | 19/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PK: Scopolamine Only, Open-label (N=13) | Efficacy: Scopolamine (Crossover, Double-blind) (N=23) | Efficacy: Placebo (Crossover, Double-blind) (N=23)
Nonserious AEs (General disorders) | 11 (42) | 18 (82) | 19 (65) — Nonserious adverse events were AEs lacking clinical significance and monitored/assessed without regard to the specific Adverse Event Term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No